CLINICAL TRIAL: NCT03512587
Title: Personalized Quantum Sonotherapy in Regional Anesthesia Peripheral Nerve Block: Randomized and Controlled Clinical Trial
Brief Title: Personalized Quantum Sonotherapy in Regional Anesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CES University (Other)
Responsible Party: Principal Investigator, Ana Sofia Arango Gutierrez, Medical Doctor, CES University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 645
Record Dates: First submitted 2018-03-25; First posted 2018-05-01 (Actual); Last update posted 2018-05-01 (Actual); Status verified 2018-04

CONDITIONS: Pain, Postoperative; Anxiety
Keywords: Personalized quantum sonotherapy; Regional anesthesia; Peripheral nerve block
MeSH Terms: conditions — Pain, Postoperative; Anxiety Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Personal quantum sonotherapy group (Experimental): Patients who will listen through MP3 devices the personalized quantum sonotherapy previously created through a especialized software, before the application of regional anesthesia.
  Interventions: Procedure: Personalized quantum sonotherapy
- Control group (Placebo Comparator): Patients will wear headphones but without playing the personalized quantum sonotherapy
  Interventions: Procedure: Placebo

INTERVENTIONS:
Procedure: Personalized quantum sonotherapy — Quantum sonotherapy is an alternative non-pharmacological treatment that effects a molecular reorganization that occurs after the sound stimulus. The audible words and their waves have the ability to generate vibrations and stimulate the psycho-neuro-endocrine chain, independent of the semantic meaning of the words. It is an alternative therapy that uses non-musical sound waves.
  Arms: Personal quantum sonotherapy group
Procedure: Placebo — Headphones will be place in patients without playing quantum sonotherapy
  Arms: Control group

SUMMARY:
The objetive of the study is to evaluate the effect of personalized quantum sonotherapy on the level of anxiety and pain in outpatients schedule for orthopedic surgery under regional anesthesia in a second level center. The investigators believed that personalized quantum sonotherapy could reduce the levels of anxiety and pain before and after surgery evaluated through hemodynamic variables and scales for pain (analogous visual scale) and anxiety (STAI Spielberger anxious state questionnaire).

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for elective orthopedic ambulatory surgery under regional anesthesia
* Age between 18 and 60 years.
* Patients with anesthetic risk ASA 1 and 2.
* Patients without contraindications for the administration of opioids and benzodiazepines.
* Patients living in the metropolitan area who have a telephone line and can be contacted by telephone within the first 48 hours through calls at 24 and 48 hours after surgery, made by the researchers at the number previously reported by the patient.
* Patients with an adequate level of understanding, who are able to communicate by telephone and understand a numerical scale.
* Patients who agree to participate in the work.

Exclusion Criteria:

* Patients with auditory and cognitive problems.
* Patients requiring general anesthesia at some time during the intraoperative period.
* Patients with morbid obesity.
* Patients consuming anxiolytics in the last month.
* Patients whose start of surgery is after 45 minutes of the blockade.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2017-03-31 (Actual); Study Completion 2017-03-31 (Actual)

PRIMARY OUTCOMES:
Pain | 48 hours (From the moment before surgery when the sonotherapy is apply until 48 hours after surgery)
  To assess the effect of personalized quantum sonotherapy on the level of pain of patients taken to orthopedic surgery under regional anesthesia through pain score visual analoge score (VAS). VAS ranges from 0 to 10 being 0 no pain an 10 the worst pain ever felted. It would be measured before and after placing de sonotherapy, 24 and 48 hour after surgery.
Anxiety | 48 hours (From the moment before surgery when the sonotherapy is apply until 48 hours after surgery)
  To assess the effect of personalized quantum sonotherapy on the level of anxiety of patients taken to orthopedic surgery under regional anesthesia through anxiety score Questionnaire of anxious state STAI (Spielberger). STAI is a score to meausre anxiety, it has 20 questions each one with a possible value from 0 to 3 points. Total score is evaluated adding each score for each question, and it goes from 0 to 60 points, being 60 de higest score for anxiety. It would be measured before and after placing de sonotherapy, 24 and 48 hour after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Mara P Gonzalez, MD, Principal Investigator — University CES
Locations (1):
- Instituto Colombiano del Dolor, Medellín, Antioquia, Colombia

IPD SHARING:
Plan to Share IPD: Undecided